CLINICAL TRIAL: NCT06916637
Title: Clinical Study on the Application of 18F-HER2 Affibody PET Imaging in HER2-Expressing Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Other Study IDs: QDFY-NM-25006
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Breast Cancer, HER2-Expression
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 18F-HER2 Affibody PET scan
  Interventions: Radiation: 18F-HER2 Affibody PET scan

INTERVENTIONS:
Radiation: 18F-HER2 Affibody PET scan — HER2 Affibody, labeled with PET radio-nuclide 18F will be used as a molecular imaging tracer for PET scan. All participants will undergo 18F-HER2 Affibody PET scan.

SUMMARY:
This study aims to evaluate the clinical utility of 18F-labeled HER2 Affibody PET for diagnosing and monitoring HER2-expressing breast cancer. HER2, a protein overexpressed in certain malignancies including breast cancer, serves as a critical biomarker for targeted therapies.The HER2 Affibody-an engineered 7 kDa protein with nanomolar affinity for HER2-leverages its rapid tumor penetration and clearance kinetics to achieve high-contrast PET imaging. This study aims to evaluate the diagnostic efficacy of 18F-HER2 Affibody PET in early detection, clinical staging, and treatment response monitoring, thereby providing novel imaging evidence to guide personalized therapeutic strategies for patients with HER2-expressing breast cancer.

DETAILED DESCRIPTION:
Human epidermal growth factor receptor 2 (HER2) is a transmembrane receptor protein with tyrosine kinase activity that plays a crucial role in cell growth, activation, and proliferation. While minimally expressed in normal tissues, HER2 is highly expressed in various malignant tumors, especially breast cancer, making it a key target for breast cancer diagnosis and treatment.HER2-positivity was defined with Immunohistochemistry (IHC) 3+ or IHC 2+ followed by Fluorescence In Situ Hybridization（FISH） showing HER2 amplification.HER2-low was defined IHC 1+ or IHC 2+ with negative FISH . Conventional diagnostic approaches like biopsy are inherently invasive and lack the capability for longitudinal evaluation of HER2 expression dynamics.The HER2-targeted Affibody molecule demonstrates superior diagnostic potential compared to traditional antibodies, attributed to its enhanced specificity, compact molecular structure enabling rapid biodistribution (achieving optimal blood clearance within 1-4 hours post-injection), and consequent high-contrast imaging capabilities. As a novel positron emission tomography (PET) tracer, 18F-HER2 Affibody holds promise for delivering precise, non-invasive quantification of HER2 status. This study seeks to systematically assess the diagnostic accuracy of 18F-HER2 Affibody PET in tumor staging and treatment stratification, while concurrently investigating its prognostic value through longitudinal treatment response monitoring in breast cancer patients with HER2-overexpressing tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years, ECOG score 0 or 1.
* Clinically or pathologically confirmed diagnosis of patients with HER2 expression breast cancer or suspected expression breast cancer.
* Life expectancy ≥ 12 weeks.
* At least one measurable target lesion according to RECIST 1.1 criteria.
* All participants of reproductive potential (regardless of gender) must commit to using effective contraceptive methods throughout the trial participation and for 6 months after the last PET scan.
* Ability to understand and voluntarily sign the informed consent form, with good compliance.

Exclusion Criteria:

* Severe hepatic or renal dysfunction.
* Pregnant or lactating women, or women planning to become pregnant.
* Inability to lie supine for half an hour.
* Refusal to participate in this clinical study.
* Suffering from claustrophobia or other mental illnesses.
* Other conditions that the investigator deems unsuitable for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for this clinical trial consists of adults aged 18 to 75 years with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. Participants must have a clinically or pathologically confirmed diagnosis of HER2 expression breast cancer or suspected HER2 expression breast cancer. A life expectancy of at least 12 weeks is required, along with the presence of at least one measurable target lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. All participants of reproductive potential must agree to use effective contraceptive methods throughout the trial and for six months after the last PET scan. Additionally, participants must be able to understand and voluntarily sign the informed consent form，demonstrating good compliance with the study protocol.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
SUV | 2 years
  The uptake of the tracer in the primary and metastatic tumor lesions by measuring standardized uptake value (SUV) on PET

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No